CLINICAL TRIAL: NCT06136676
Title: From the Heart Multi-Centre Study: Comparing the Effects of Spiritual and Secular Meditation on Psychophysiology, Cognition, Mental Health, and Social Functioning in Healthy Adults
Brief Title: From the Heart: Comparing the Effects of Spiritual and Secular Meditation on Psychophysiology, Cognition, Mental Health, and Social Functioning in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Collaborators: Donders Centre for Cognitive Neuroimaging (Other); Kuriakose Elias College Mannanam (Unknown); Little Flower Institute of Social Sciences and Health (LISSAH) College (Unknown)
Responsible Party: Principal Investigator, Miguel Farias, Associate Professor, Coventry University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TWCF0595; 0595 (Other Grant/Funding Number: Templeton World Charity Foundation)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Prosocial Behavior; Forgiveness; Empathy; Pain; Attention; Depression; Stress; Anxiety; Mental Well-being
Keywords: Christian spiritual meditation; Islamic spiritual meditation; Mindfulness; Prosociality; Forgiveness; Empathy; Pain; Attention; Depression; Stress; Anxiety; Well-being; Heart-centred spirituality
MeSH Terms: conditions — Altruism; Pain; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study consists of 3 arms, including:
  Arm 1 - experimental groups: Heart-Centred Spiritual Meditation. Within this arm, the interventions encompass Islamic heart-centred contemplation and Christian heart-centred contemplation. Participants allocated to the spiritual meditation groups will receive either Islamic or Christian heart-centred contemplation intervention, depending on their respective religious affiliations.
  Arm 2 - active control group: Mindfulness-based Stress Reduction. Participants assigned to the active control group will receive mindfulness intervention. This arm mirrors the time commitment and level of engagement of the contemplation interventions.
  Arm 3 - passive control group: Waitlist control. Participants assigned to the waitlist control group will not receive any intervention.
Who Masked: Outcomes Assessor
Masking Description: Blinded data analysis. The researcher who analyzes the data will be kept unaware of the information about the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heart-centred spiritual meditation (Experimental): Intervention 1: Christian contemplation and Intervention 2: Islamic contemplation
  Interventions: Behavioral: Arm 1 - Heart-Centred Spiritual Meditation: Christian contemplation; Behavioral: Arm 1 - Heart-Centred Spiritual Meditation: Islamic contemplation
- Mindfulness Meditation (MBRS) (Active Comparator): Intervention 3: Mindfulness Meditation (MBRS)
  Interventions: Behavioral: Arm 2 - Action Control: Mindfulness Meditation
- Waitlist control (No Intervention): No Intervention: Participants in this condition will not receive any intervention and the outcome measures will be only collected at time points T1 and T2. After T2 testing, they will be given access to either the Christian or Islamic intervention.

INTERVENTIONS:
Behavioral: Arm 1 - Heart-Centred Spiritual Meditation: Christian contemplation — Participants assigned to this condition will receive daily audio instructions of approximately 20 minutes daily over the course of 8 weeks focused on Christian contemplation delivered through a mobile app. The intervention will consist of a core contemplative practice focused on heart visualisation based on Christian tradition and prayer recitation with breathing to focus their attention on and connection to God.
  Arms: Heart-centred spiritual meditation
Behavioral: Arm 1 - Heart-Centred Spiritual Meditation: Islamic contemplation — Participants assigned to this condition will receive daily audio instructions of approximately 20 minutes daily over the course of 8 weeks, focused on Islamic contemplation delivered through a mobile app. The intervention will consist of a core contemplative practice focused on heart visualisation based on Islamic tradition and prayer recitation with breathing to focus attention on and connection to God.
  Arms: Heart-centred spiritual meditation
Behavioral: Arm 2 - Action Control: Mindfulness Meditation — Participants assigned to this condition will receive daily audio instructions of approximately 20 minutes daily over the course of 8 week, focused on mindfulness meditation delivered through a mobile app. The intervention will consist of the mindfulness-based stress reduction program which emphasizes focused attention on breathing and sensations as well as the practice of non-judgemental acceptance of the present experience.
  Arms: Mindfulness Meditation (MBRS)

SUMMARY:
The purpose of this study is to investigate and compare the effects of Christian and Islamic heart-centred spiritual meditation to mindfulness meditation and waitlist control conditions, respectively, in healthy adults. The potential effects will be studied at multiple levels, with a focus on psychophysiology, cognition, mental health, and social functioning.

DETAILED DESCRIPTION:
Background

Secular forms of meditation have been widely accepted as an effective tool to promote well-being and as therapeutic strategies. The popularity of such practices, most notably mindfulness meditation, can be attributed to the substantial body of research on their beneficial effects in the past few decades. While these practices are loosely based on Eastern traditions, and actively reduce emotional reactivity, some Western spiritual meditations have retained their God-centred focus and aim to elicit strong emotions. The current study aims to examine the effects of heart-centred contemplation based on Christian and Islamic traditions on mental, physical, cognitive, and social well-being, compare the outcomes of these exercises to mindfulness meditation, and investigate the external correlates of the outcomes.

Aims

The present study aims to recruit healthy adults to investigate and compare the effects of Christian and Islamic heart-centred spiritual meditation to mindfulness meditation (Mindfulness-based stress reduction; MBSR) and waitlist control, respectively. The potential effects will be examined using measures from multiple domains, with a focus on psychophysiology, cognition, mental health, and social functioning. Additionally, the study aims to examine the possible external correlates of the outcomes by testing perspective-taking, affect, religiosity, spiritual experiences, closeness to God, closeness to the offender, and credibility/expectancies about the spiritual meditation program. The study seeks to understand the impact of different types of meditation practices on the well-being of individuals.

Participants

This study will apply a mixed method repeated measures design to examine a three-arm stratified randomised control trial with healthy samples of Christians and Muslims in multiple testing centres in India. Assessments will be conducted at three time points: pre-intervention (T1), after intervention (T2), and at a 3-month follow-up (T3). Eligible participants will be first stratified into Christian and Islamic samples and then randomly allocated to one of the three conditions: religious contemplation (either Christian or Islamic spiritual meditation based on their religions), mindfulness meditation, or waitlist control.

Administration of intervention

The intervention will consist of an 8-week app-based program, including approximately 20-minute daily audio-guided instructions of either one of the spiritual meditations or mindfulness meditation. Participants from the waitlist control will not receive any intervention, but they will be given access to Christian or Islamic meditation app after the experiment is completed.

Outcome measures

Outcome measures consist of domains related to interpersonal functioning, physiology, attention, mental health, spirituality.

Primary outcomes will be the interpersonal functioning domain including measures of prosociality, forgiveness, empathy, and perspective taking.

Secondary outcomes include domains concerning physiology, attention, and mental health. Physiology domain encompasses pain tolerance, pain intensity, stress reactivity (heart rate and heart rate variability), psychophysiological reactivity associated with forgiveness (heart rate and heart rate variability). Attention domain includes measures of alerting attention, orienting attention, and executive attention networks. Mental health domain involves self-reported stress, depression, anxiety, subjective well-being, and positive and negative affect.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* able to read, speak and understand English
* willing to be randomly assigned to all the conditions, with religious affiliation restricting allocation to either the Christian or Islamic type of spiritual meditation conditions
* consider oneself to be a Christian or Muslim and pray at least weekly

Exclusion Criteria:

* currently suffer from any mental health conditions or use medication to manage mental health conditions
* long-term serious physical medical problems, such as liver, brain, kidney, or other life-threatening chronic diseases
* a history of a heart condition, high blood pressure, Raynaud syndrome, diabetes, or musculoskeletal condition
* the current use of anxiolytics/mood stabilizers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Interpersonal functioning: Change in Prosociality (1) | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  The number of game points (0-10) that a participant is willing to allocate to another individual as measured by the Dictator Game
Interpersonal functioning: Change in Prosociality (2) | Pre-intervention (collected up to 1 week before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Social value orientation scores as measured by the social value orientation slider measure. The higher scores represent greater prosocial preferences while lower scores represent greater self-interest preferences
Interpersonal functioning: Change in Prosociality (3) | Post-intervention (collected up to two weeks after the 8-week intervention)
  The percentage of compensation fees that participants are willing to donate to a charity
Interpersonal functioning: Changes in self-reported Forgiveness | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  A self-reported forgiveness scale assessed within a forgiveness task, ranging from 0 (Not at all) to 20 (Completely). High scores reflect a higher level of forgiveness, while lower scores indicate a lower level of forgiveness
Interpersonal functioning: Changes in self-reported Empathy | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  A self-reported empathy scale assessed within a forgiveness task, ranging from 0 (Not at all) to 20 (Completely). High scores reflect a higher level of empathy, while lower scores indicate a lower level of empathy.
Interpersonal functioning: Change in Perspective Taking | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  Interpersonal Reactivity Index (IRI) - Perspective Taking scale. The 7-item Perspective Taking scale from IRI measures one's tendency to take the point of view of others. Participants are asked to rate how closely the statements describe them on a 5-point Likert scale ranging from A (Does not describe me well) to E (Describes me very well). The total scores range from 0 - 28. Higher scores indicate greater perspective-taking

SECONDARY OUTCOMES:
Physiology: Change in Pain Tolerance | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  The duration (in seconds) that a participant endures painful stimulation assessed during an endurance task
Physiology: Change in Pain Intensity | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  0-10 Numerical Rating Scale
Physiology: Change in Stress Reactivity (1) | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Heart rate
Physiology: Change in Stress Reactivity (2) | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Heart rate variability
Physiology: Change in psychophysiological reactivity associated with forgiveness (1) | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Heart rate assessed during a forgiveness task.
Physiology: Change in psychophysiological reactivity associated with forgiveness (2) | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Heart rate variability assessed during a forgiveness task
Attention: Change in Alerting Attention network | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Reaction time assessed through a 10-minute version of Attentional Network Task (CRSD-ANT)
Attention: Change in Orienting Attention network | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Reaction time assessed through a 10-minute version of Attentional Network Task (CRSD-ANT)
Attention: Change in Executive Attention network | Pre-intervention (collected up to 3 hours before the intervention), and post-intervention (collected up to two weeks after the 8-week intervention)
  Reaction time assessed through a 10-minute version of Attentional Network Task (CRSD-ANT)
Mental health: Change in self-reported Stress | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a 21-item self-report questionnaire that comprises three distinct subscales: depression, anxiety, and stress, with each containing 7 items. Participants are asked to rate the extent of the statements applied to them over the past week using a 4-point rating scale, ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). Higher scores on stress scale reflect a greater severity of the stress symptoms, whereas lower scores indicate a milder experience of these symptoms
Mental health: Change in self-reported Depression | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21): Depression subscale, ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). Higher scores on depression scale reflect a greater severity of the depression symptoms, whereas lower scores indicate a milder experience of these symptoms
Mental health: Change in self-reported Anxiety | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21): Anxiety subscale, ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). Higher scores on anxiety scale reflect a greater severity of the anxiety symptoms, whereas lower scores indicate a milder experience of these symptoms
Mental health: Change in Subjective Wellbeing | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  Well-Being Index (WHO-5). WHO-5 is a 5-item self-report questionnaire measuring subjective wellbeing. Participants are asked to rate their feelings in the past 2 weeks using a 6-Likert scale, ranging from 0 (At no time) to 5 (All of the time). The raw score is multiplied by 4 and the final scores range from 0-100. A score of 0 indicates the lowest possible level of wellbeing, whereas a score of 100 reflects the highest possible level of wellbeing
Mental health: Change in self-report Positive and Negative Affect (1) | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  International Positive and Negative Affect Schedule (PANAS) Short Form (I-PANAS-SF). I-PANAS-SF is a 10-item self-report questionnaire measuring 5 items of positive affect and 5 items of negative affect. Participants are asked to rate their general feelings and emotions on a 5-point Likert scale ranging from 1 (Never) to 5 (Always). Higher scores indicate a greater level of positive affect, and lower scores represent a lower level of negative affect
Mental health: Change in self-report Positive and Negative Affect (2) | Throughout the 8 weeks intervention
  5-item Smiley Face Likert scale within the meditation app. The scale assesses participants' feelings before and after their daily contemplative / mindfulness practices. Participants are asked to choose one out of the five emoji faces on the scale to indicate their current feelings ranging from a very sad face to a very happy face

OTHER OUTCOMES:
Spirituality: Change in Spiritual Experiences | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  The Daily Spiritual Experience Scale (DSES). DSES is a 16-item self-report questionnaire. Participants are asked to rate their daily spiritual experiences. 15 items are rated on a 6-point Likert scale from 1 (Many times a day) to 6 (Never or almost never) and 1 item is rated on a 4-point Likert scale from 1 (Not close) to 4 (As close as possible). Higher scores indicate greater spirituality
Spirituality: Change in Closeness to God | Pre-intervention (collected up to 1 week before the intervention), post-intervention (collected up to 2 weeks after the 8-week intervention), and at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  Inclusion-of-God-in-the-self scale (adapted from Inclusions of Others in Self scale). The scale consists of 7 pairs of pictorial circles with one circle of each pair being labelled as Self, and the other circle being labelled as God. Participants are asked to choose 1 of the 7 pairs of circles that best describes their relationship with God. The pairs of circles have different degrees of overlap, ranging from the 1st pair (no overlap) to the 7th pair (most overlap). The greater the overlap in the circles corresponds to a closer relationship with God
Spirituality: Religiosity | Pre-intervention (collected up to 1 week before the intervention)
  Duke University Religiosity Index (DUREL). DUREL is a 5-item self-report questionnaire measuring three major dimensions of religious involvement with three subscales: organizational religious activity (ORA), non-organizational religious activity (NORA), and intrinsic religiosity (IR). Participants are asked to rate their religious involvement (ORA and NORA) on a 6-point Likert scale ranging from 1 (Never) to 6 (More than once a week/day) and rate their religious beliefs or experience (IR) on a 5-point Likert scale ranging from 1 (Definitely not true) to 5 (Definitely true of me). Higher scores indicate a higher religiosity
Credibility/Expectancy of the meditation practices | Pre-intervention (collected up to 1 week before the intervention)
  Credibility/Expectancy questionnaire. This is a 4-item self-report questionnaire that assesses participants' beliefs about the efficacy and credibility of the contemplative practices on a 9-point Likert scale from 1 (Not at all) to 9 (Very much). Higher scores indicate greater positive expectancies
Closeness to the offender | Pre-intervention (collected up to 3 hours before the intervention)
  The Inclusion-of-Other-in-the-Self scale assessed within the forgiveness task. It is a pictorial scale consists of seven pairs of circles, with one circle of each pair labelled as Self and the other circle labelled as Other. Participants are asked to choose the pair of circles that best describes their relationship with the offender. The pairs of circles have different degrees of overlap, ranging from the 1st pair (no overlap) to the 7th pair (most overlap). The greater the overlap in the circles, the closer the relationship with the offender
Demographics: Age | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Demographics: Ethnicity | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Demographics: Gender Identity | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Demographics: Biological Sex | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Socioeconomic Status: Employment status | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Socioeconomic Status: Education level | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Socioeconomic Status: Annual household income | Pre-intervention (collected up to 1 week before the intervention)
  Self-report assessment
Potential adverse events in the meditative practices | Post-intervention (collected up to two weeks after the 8-week intervention)
  Self-report unpleasant events and harm questionnaire. The questionnaire is a self-report measure to assess the unpleasant events and harm in contemplative or mindfulness practices. It includes Likert ratings and free-text questions about unpleasant feelings and the harm that participants may have experienced during the contemplation or mindfulness practices
Experiences of the App-based exercises | Post-intervention (collected up to two weeks after the 8-week intervention) and at 3-month follow-up (collected up to 2 weeks following 3 months after the intervention)
  Self-report assessment about participant's experiences with the App-based exercises
Frequency of the contemplative or mindfulness practices after the end of the intervention | at 3-month follow-up (collected up to 2 weeks following 3 months after the end of the intervention)
  Self-report assessment about frequency of participant's practices after the end of the 8-week intervention
Qualitative assessment: Themes emerging from participant's meditation diary | Throughout the 8 weeks intervention
  Key themes that emerge from participants' diaries for their reflection on their experiences of the daily meditative practices
Qualitative assessment: Themes emerging from participant's daily meditative experiences | Throughout the 8 weeks intervention
  Key themes that emerge from participants' daily meditative experiences assessed within the App

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Little Flower Institute of Social Sciences and Health (LISSAH) college, Calicut, Kerala
  - Kuriakose Elias College Mannanam, Kottayam, Kerala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ainsworth B, Eddershaw R, Meron D, Baldwin DS, Garner M. The effect of focused attention and open monitoring meditation on attention network function in healthy volunteers. Psychiatry Res. 2013 Dec 30;210(3):1226-31. doi: 10.1016/j.psychres.2013.09.002. Epub 2013 Oct 14. PMID 24135553
- [Background] Aron A, Aron EN, Smollan D. Inclusion of Other in the Self Scale and the structure of interpersonal closeness. Journal of Personality and Social Psychology. 1992; 63(4): 596-612.
- [Background] Baer R, Crane C, Montero-Marin J, Phillips A, Taylor L, Tickell A, Kuyken W; MYRIAD team. Frequency of Self-reported Unpleasant Events and Harm in a Mindfulness-Based Program in Two General Population Samples. Mindfulness (N Y). 2021;12(3):763-774. doi: 10.1007/s12671-020-01547-8. Epub 2020 Dec 2. PMID 33747251
- [Background] Baesler EM, Derlega VJ, Winstead BA, Barbee A. Prayer as Interpersonal Coping in the Lives of Mothers with HIV. Communication & Theatre Arts Faculty Publications. 2003; 26(3-4): 283-295.
- [Background] Bandura A. On the psychosocial impact and mechanisms of spiritual modeling. The International Journal for the Psychology of Religion. 2003; 13(3): 167-174.
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology. 2006; 3(2): 77-101.
- [Background] Bryant RA, Marosszeky JE, Crooks J, Gurka JA. Elevated resting heart rate as a predictor of posttraumatic stress disorder after severe traumatic brain injury. Psychosom Med. 2004 Sep-Oct;66(5):760-1. doi: 10.1097/01.psy.0000138121.13198.84. PMID 15385703
- [Background] Buric I, Brazil IA, van Mulukom V. Individual differences in meditation outcomes. The Oxford Handbook of Meditation. Oxford University Press. 2021; 503-524.
- [Background] Buric I, Farias M, Jong J, Mee C, Brazil IA. What Is the Molecular Signature of Mind-Body Interventions? A Systematic Review of Gene Expression Changes Induced by Meditation and Related Practices. Front Immunol. 2017 Jun 16;8:670. doi: 10.3389/fimmu.2017.00670. eCollection 2017. PMID 28670311
- [Background] Carlson CA, Bacaseta PE, Simanton DA. A controlled evaluation of devotional meditation and progressive relaxation. Journal of Psychology and Theology. 1988; 16(4): 362-368.
- [Background] Carmo Silva C. The Phenomenology of Meditation: Commonalities and Divergences between Christian Meditation and Hindu Dhyāna. The Oxford Handbook of Meditation. Oxford University Press. 2021; 384-400.
- [Background] Charles SJ, Farias M, van Mulukom V, Saraswati A, Dein S, Watts F, Dunbar RIM. Blocking mu-opioid receptors inhibits social bonding in rituals. Biol Lett. 2020 Oct;16(10):20200485. doi: 10.1098/rsbl.2020.0485. Epub 2020 Oct 14. PMID 33050833
- [Background] Charles SJ, van Mulukom V, Brown JE, Watts F, Dunbar RIM, Farias M. United on Sunday: The effects of secular rituals on social bonding and affect. PLoS One. 2021 Jan 27;16(1):e0242546. doi: 10.1371/journal.pone.0242546. eCollection 2021. PMID 33503054
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Collicutt J, Bretherton R, Brickman J. Being Mindful, Being Christian: A guide to mindful discipleship. Monarch Book. 2016.
- [Background] Condon P, DeSteno D. Enhancing compassion: Social psychological perspectives. The Oxford Handbook of Compassion Science. Oxford University Press. 2017.
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Creswell JD, Pacilio LE, Lindsay EK, Brown KW. Brief mindfulness meditation training alters psychological and neuroendocrine responses to social evaluative stress. Psychoneuroendocrinology. 2014 Jun;44:1-12. doi: 10.1016/j.psyneuen.2014.02.007. Epub 2014 Feb 23. PMID 24767614
- [Background] Davis M. Measuring individual differences in empathy: Evidence for a multidimensional approach. Journal of Personality and Social Psychology. 1983; 44(1): 113-126.
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Farias M, Maraldi E, Wallenkampf KC, Lucchetti G. Adverse events in meditation practices and meditation-based therapies: a systematic review. Acta Psychiatr Scand. 2020 Nov;142(5):374-393. doi: 10.1111/acps.13225. Epub 2020 Aug 21. PMID 32820538
- [Background] Farias M, van Mulukom V, Kahane G, Kreplin U, Joyce A, Soares P, Oviedo L, Hernu M, Rokita K, Savulescu J, Mottonen R. Supernatural Belief Is Not Modulated by Intuitive Thinking Style or Cognitive Inhibition. Sci Rep. 2017 Nov 8;7(1):15100. doi: 10.1038/s41598-017-14090-9. PMID 29118434
- [Background] Farias M, Wikholm C. The Buddha Pill: Can Meditation Change You? Watkins. 2019.
- [Background] Farias M, Brazier D, Lalljee M. Introduction: Understanding and Studying Meditation. The Oxford Handbook of Meditation. Oxford University Press. 2021; 2-17.
- [Background] Ferreira-Valente A, Van Dyke BP, Day MA, Teotonio do Carmo C, Pais-Ribeiro J, Pimenta F, Costa RM, Jensen MP. Immediate Effects of Hypnosis, Mindfulness Meditation, and Prayer on Cold Pressor Outcomes: A Four-Arm Parallel Experimental Study. J Pain Res. 2022 Dec 23;15:4077-4096. doi: 10.2147/JPR.S388082. eCollection 2022. PMID 36582659
- [Background] Forsythe R, Horowitz JL, Savin N, Sefton M . Fairness in Simple Bargaining Experiments. Games and Economic Behavior. 1994b; 6(3): 347-369.
- [Background] Fox K, Cahn R. Meditation and the brain in health and in disease. The Oxford Handbook of Meditation. Oxford University Press. 2021.
- [Background] Fredrickson BL. Positive Emotions Broaden and Build. Advances in Experimental Social Psychology. 2013; 47: 1-53
- [Background] Goyal M, Rusch H. Mindfulness-based interventions in the treatment of physical conditions. The Oxford Handbook of Meditation. Oxford University Press. 2021; 1-25
- [Background] Guroglu B, van den Bos W, Crone EA. Fairness considerations: increasing understanding of intentionality during adolescence. J Exp Child Psychol. 2009 Dec;104(4):398-409. doi: 10.1016/j.jecp.2009.07.002. Epub 2009 Aug 11. PMID 19674756
- [Background] Hines EA, Brown GE . The cold pressor test for measuring the reactibility of the blood pressure: Data concerning 571 normal and hypertensive subjects. American Heart Journal. 1936; 11(1): 1-9.
- [Background] Hisham AR. Towards a systematic Qura'nic theory of personality. Mental Health, Religion & Culture. 2012; 15(3): 217-233.
- [Background] Kabat-Zinn J. Mindfulness-based interventions in context: Past, present, and future. Clinical Psychology: Science and Practice. 2003; 10(2): 144-156.
- [Background] Kabat-Zin J. Full Catastrophe Living: Using the Wisdom of Your Body and Mind to Face Stress, Pain, and Illness. Penguin Random House. 2013.
- [Background] Karremans JC, van Schie HT, van Dongen I, Kappen G, Mori G, van As S, Ten Bokkel IM, van der Wal RC. Is mindfulness associated with interpersonal forgiveness? Emotion. 2020 Mar;20(2):296-310. doi: 10.1037/emo0000552. Epub 2019 Jan 17. PMID 30652883
- [Background] Kemeny ME, Foltz C, Cavanagh JF, Cullen M, Giese-Davis J, Jennings P, Rosenberg EL, Gillath O, Shaver PR, Wallace BA, Ekman P. Contemplative/emotion training reduces negative emotional behavior and promotes prosocial responses. Emotion. 2012 Apr;12(2):338-50. doi: 10.1037/a0026118. Epub 2011 Dec 12. PMID 22148989
- [Background] Kemp AH, Brunoni AR, Santos IS, Nunes MA, Dantas EM, Carvalho de Figueiredo R, Pereira AC, Ribeiro AL, Mill JG, Andreao RV, Thayer JF, Bensenor IM, Lotufo PA. Effects of depression, anxiety, comorbidity, and antidepressants on resting-state heart rate and its variability: an ELSA-Brasil cohort baseline study. Am J Psychiatry. 2014 Dec 1;171(12):1328-34. doi: 10.1176/appi.ajp.2014.13121605. Epub 2014 Oct 31. PMID 25158141
- [Background] Koenig HG, McCullough ME, Larson DB. Handbook of Religion and Health. Oxford University Press. 2001.
- [Background] Koenig HG, Büssing A .The Duke University Religion Index (DUREL): A Five-Item Measure for Use in Epidemological Studies. Religions. 2010, 1(1): 78-85.
- [Background] Kreplin U, Farias M, Brazil IA. The limited prosocial effects of meditation: A systematic review and meta-analysis. Sci Rep. 2018 Feb 5;8(1):2403. doi: 10.1038/s41598-018-20299-z. PMID 29402955
- [Background] Kuczok M. The Interplay of Metaphor and Metonymy in Christian Symbols. Metaphor and Symbol. 2020; 35(4): 236-249.
- [Background] Kuggle S. The Brilliance of Hearts. Islam in South Asia in Practice. Princeton University Press. 2010.
- [Background] Laird M. Into the Silent Land: A Guide to the Christian Practice of Contemplation. Oxford University Press. 2006.
- [Background] Marchant J. Cure: A Journey into the Science of Mind Over Body. Two Ravens Press. 2016.
- [Background] May RW, Cooper AN, Fincham FD. Prayer in Marriage to Improve Wellness: Relationship Quality and Cardiovascular Functioning. J Relig Health. 2020 Dec;59(6):2990-3003. doi: 10.1007/s10943-019-00829-3. PMID 31065881
- [Background] Morgan D. The Sacred Heart of Jesus: The Visual Evolution of a Devotion. Amsterdam University Press. 2008.
- [Background] Murphy RO, Ackermann KA, Handgraaf M. Measuring social value orientation. Judgment and Decision Making. 2011; 6(8): 771-781.
- [Background] Oman D. Studying the effects of meditation: The first fifty years. The Oxford Handbook of Meditation. Oxford University Press. 2021.
- [Background] Oman D, Hedberg J, Thoresen CE. Passage meditation reduces perceived stress in health professionals: a randomized, controlled trial. J Consult Clin Psychol. 2006 Aug;74(4):714-9. doi: 10.1037/0022-006X.74.4.714. PMID 16881779
- [Background] Pargament KI. The Psychology of Religion and Coping: Theory, Research, and Practice. New York: Guilford Press. 1997.
- [Background] Parrott, J. How to be a Mindful Muslim: An Exercise in Islamic Meditation. Yaqeen Institute for Islamic Research. 2017.
- [Background] Porcelli AJ. An alternative to the traditional cold pressor test: the cold pressor arm wrap. J Vis Exp. 2014 Jan 16;(83):e50849. doi: 10.3791/50849. PMID 24457998
- [Background] Saab PG, Llabre MM, Hurwitz BE, Schneiderman N, Wohlgemuth W, Durel LA, Massie C, Nagel J. The cold pressor test: vascular and myocardial response patterns and their stability. Psychophysiology. 1993 Jul;30(4):366-73. doi: 10.1111/j.1469-8986.1993.tb02058.x. PMID 8327622
- [Background] Sanfey AG. Social decision-making: insights from game theory and neuroscience. Science. 2007 Oct 26;318(5850):598-602. doi: 10.1126/science.1142996. PMID 17962552
- [Background] Sedlmeier P, Eberth J, Schwarz M, Zimmermann D, Haarig F, Jaeger S, Kunze S. The psychological effects of meditation: a meta-analysis. Psychol Bull. 2012 Nov;138(6):1139-71. doi: 10.1037/a0028168. Epub 2012 May 14. PMID 22582738
- [Background] Shalev AY, Sahar T, Freedman S, Peri T, Glick N, Brandes D, Orr SP, Pitman RK. A prospective study of heart rate response following trauma and the subsequent development of posttraumatic stress disorder. Arch Gen Psychiatry. 1998 Jun;55(6):553-9. doi: 10.1001/archpsyc.55.6.553. PMID 9633675
- [Background] Shapiro D, Walsh R. Meditation: Classic and contemporary perspectives. Aldine. 1984.
- [Background] Skwara A, King B, Saron C. Studies of training compassion: What have we learned; what remains unknown? Oxford Handbook of Compassion Science. Oxford University Press. 2017.
- [Background] Spearing AC. The Cloud of Unknowing and Other Works (Penguin Classics). Penguin Books Ltd. 2001.
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA. Manual for the State-Trait Anxiety Inventory. CA: Consulting Psychologists Press. 1983.
- [Background] Tang YY, Bruya B. Mechanisms of Mind-Body Interaction and Optimal Performance. Front Psychol. 2017 May 9;8:647. doi: 10.3389/fpsyg.2017.00647. eCollection 2017. No abstract available. PMID 28536540
- [Background] Tang YY, Ma Y, Wang J, Fan Y, Feng S, Lu Q, Yu Q, Sui D, Rothbart MK, Fan M, Posner MI. Short-term meditation training improves attention and self-regulation. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17152-6. doi: 10.1073/pnas.0707678104. Epub 2007 Oct 11. PMID 17940025
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Underwood LG. The Daily Spiritual Experience Scale: Overview and Results. Religions, 2011; 2(1): 29-50.
- [Background] Van Cappellen P, Toth-Gauthier M, Saroglou V, Fredrickson BL. Religion and Well-Being: The Mediating Role of Positive Emotions. Journal of Happiness Studies. 2014; 17(2): 485-505.
- [Background] Van Dam NT, van Vugt MK, Vago DR, Schmalzl L, Saron CD, Olendzki A, Meissner T, Lazar SW, Kerr CE, Gorchov J, Fox KCR, Field BA, Britton WB, Brefczynski-Lewis JA, Meyer DE. Mind the Hype: A Critical Evaluation and Prescriptive Agenda for Research on Mindfulness and Meditation. Perspect Psychol Sci. 2018 Jan;13(1):36-61. doi: 10.1177/1745691617709589. Epub 2017 Oct 10. PMID 29016274
- [Background] vanOyen Witvliet C, Ludwig TE, Vander Laan KL. Granting forgiveness or harboring grudges: implications for emotion, physiology, and health. Psychol Sci. 2001 Mar;12(2):117-23. doi: 10.1111/1467-9280.00320. PMID 11340919
- [Background] Visted E, Vøllestad J, Nielsen MB, Nielsen GH. The Impact of Group-Based Mindfulness Training on Self-Reported Mindfulness: a Systematic Review and Meta-analysis. Mindfulness. 2014; 6(3): 501-522.
- [Background] Wachholtz AB, Malone CD, Pargament KI. Effect of Different Meditation Types on Migraine Headache Medication Use. Behav Med. 2017 Jan-Mar;43(1):1-8. doi: 10.1080/08964289.2015.1024601. Epub 2015 Apr 11. PMID 25864906
- [Background] Wachholtz AB, Pargament KI. Is spirituality a critical ingredient of meditation? Comparing the effects of spiritual meditation, secular meditation, and relaxation on spiritual, psychological, cardiac, and pain outcomes. J Behav Med. 2005 Aug;28(4):369-84. doi: 10.1007/s10865-005-9008-5. PMID 16049627
- [Background] Ware K. How do we enter the heart? Paths to the Heart: Sufism and the Christian East. Bloomington, Indiana: World Wisdom. 2002; 2-23.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Weaver B, Bedard M, McAuliffe J. Evaluation of a 10-minute version of the Attention Network Test. Clin Neuropsychol. 2013;27(8):1281-99. doi: 10.1080/13854046.2013.851741. Epub 2013 Nov 9. PMID 24205860
- [Background] Wiech K, Farias M, Kahane G, Shackel N, Tiede W, Tracey I. An fMRI study measuring analgesia enhanced by religion as a belief system. Pain. 2008 Oct 15;139(2):467-476. doi: 10.1016/j.pain.2008.07.030. Epub 2008 Sep 5. PMID 18774224
- [Background] Williams JM, Crane C, Barnhofer T, Brennan K, Duggan DS, Fennell MJ, Hackmann A, Krusche A, Muse K, Von Rohr IR, Shah D, Crane RS, Eames C, Jones M, Radford S, Silverton S, Sun Y, Weatherley-Jones E, Whitaker CJ, Russell D, Russell IT. Mindfulness-based cognitive therapy for preventing relapse in recurrent depression: a randomized dismantling trial. J Consult Clin Psychol. 2014 Apr;82(2):275-86. doi: 10.1037/a0035036. Epub 2013 Dec 2. PMID 24294837
- [Background] Yazaki S. Islamic Mysticism and Abu Talib Al-Makki: The Role of the Heart. Routledge. 2013.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Lovibond SH, Lovibond PF. Manual for the Depression Anxiety Stress Scales. Psychology Foundation: Sydney, Australia. 1995.
- [Derived] Ng CF, Farias M, Brazil IA. Interpersonal and individual effects of an app-based Christian and Islamic heart meditation intervention in healthy adults: protocol of a stratified randomised controlled trial. BMC Psychol. 2024 Sep 27;12(1):509. doi: 10.1186/s40359-024-02022-y. PMID 39334310